CLINICAL TRIAL: NCT07271381
Title: THREAT: Testing Harms Related to Exposure to Allergenic and Epithelial Toxins
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 10002257; 002257-I
Record Dates: First submitted 2025-12-06; First posted 2025-12-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12-03

CONDITIONS: Allergic; Inflammatory
Keywords: Environmental Exposures; Skin barrier dysfunction; Skin impedance
MeSH Terms: interventions — Environmental Exposure

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Common Airway (Experimental): Exposure to a sham air purifier, and wall art with foam and polyurethane.
  Interventions: Other: Environmental Exposures
- Common Gastrointestinal (Experimental): Exposure to an ultra processed diet.
  Interventions: Other: Environmental Exposures
- Common Skin (Experimental): Exposure to toothpaste, body wash, shampoo, and detergents containing sodium lauryl sulfate and other hazardous agents (commonly used likely toxic ingredients).
  Interventions: Other: Environmental Exposures
- Pure Airway (Other): Exposure to wall art without foam and polyurethane.
  Interventions: Other: Control Exposures
- Pure Gastrointestinal (Other): Exposure to a a minimally processed diet.
  Interventions: Other: Control Exposures
- Pure Skin (Other): Exposure to SLS-free and toxin free toothpaste, body wash, shampoo, detergents, non-synthetic clothing, and sheets.
  Interventions: Other: Control Exposures

INTERVENTIONS:
Other: Environmental Exposures — Toothpaste, skin lotion, hand soap, body wash, laundry detergent, shampoo containing sodium lauryl sulfate (SLS), wall art with foam and polyurethane, and processed food.
  Arms: Common Airway; Common Gastrointestinal; Common Skin
Other: Control Exposures — SLS-free, toxin free toothpaste, body wash, shampoo, detergents, non-synthetic clothing, and sheets, a minimally processed diet, and wall art without foam and polyurethane.
  Arms: Pure Airway; Pure Gastrointestinal; Pure Skin

SUMMARY:
Background:

Allergic and inflammatory conditions have been increasing over the years. Many factors may play a role in this. Every day, people are exposed to pollution and chemicals in our foods, clothing, and all of the cleaning, hygiene, and other products we use. Studies have suggested there may be links between these environmental exposures and allergic and inflammatory illnesses. Researchers want to know more about how these exposures affect our health.

Objective:

To learn how everyday exposure to common substances affects people s health.

Eligibility:

Healthy people aged 18 to 80 years.

Design:

Participants will have 2 stays in the hospital. Each stay will last 7 days, and the stays will be spaced 4 to 6 weeks apart. During both stays, participants will remain confined to their room. They will eat only food from the menu, and they will use only provided products for personal care. (They may bring their own electronic devices, such as their phone and computer.)

One stay will be in a pure room. Participants will breathe filtered air, eat unprocessed foods, and use personal care products with fewer chemicals.

One stay will be in a room that allows exposure to common environmental chemicals. Some participants will be limited to only 1 type of exposure: chemicals thought to affect only skin, gut, or respiratory health. Some participants will be exposed to all 3 types.

Participants will undergo testing. Blood, skin cell, urine, mouth swabs, and stool samples will be taken. They will have lung tests, smell tests, and tests that measure the health of their skin.

These tests will be repeated in outpatient visits 2 weeks after each hospital stay....

DETAILED DESCRIPTION:
Study Description:

In this study, we aim to investigate whether there is a link between lifestyle exposures, inflammation, and disease by exposing participants to environments with real-world levels of common skin and hair products (eg, soaps, shampoos), a typical Western diet of processed food, and/or ubiquitous air exposures, and to environments with cleaner, more natural contactants and less processed food. Participants will spend up to 7 days as an inpatient in a controlled environment with the assigned exposures, and up to 7 days as an inpatient in a cleaner environment. We will collect a variety of biospecimens and data throughout the inpatient stays to identify changes in skin, gastrointestinal (GI), and airway survey parameters.

The study will consist of 2 stages with a crossover design in each stage. Stage 1 will be divided into 3 cohorts: one cohort to identify changes in skin, one for GI changes, and one for airway changes. Within each cohort, participants will be block randomized to spend up to 7 days in the inpatient unit with either the specifically assigned experimental (common) or control (pure) exposures. Within each of the 3 cohorts, the common exposures will target a specific organ system (skin, GI, or airway). After a brief washout period, participants will then crossover to the other targeted exposure (ie, from common to pure or vice versa), for an additional inpatient stay of up to 7 days. The findings from each participant s first inpatient stay will be compared to findings from their crossover second inpatient stay.

The data collected from Stage 1 may be used to clarify the survey parameters of participants enrolled into Stage 2, in which new participants will be randomized to all common exposure domains (skin + GI + airway) vs. pure (control) and then a crossover.

Objectives:

Stage 1 Primary Objectives:

1. Cohort 1: Determine the effects of common vs. pure exposures on the skin in healthy volunteers.
2. Cohort 2: Determine the effects of common vs. pure exposures on the GI tract in healthy volunteers.
3. Cohort 3: Determine the effects of common vs. pure exposures on the airway in healthy volunteers.

Stage 1 Secondary Objective: Determine the combined effects of common vs. pure exposures on the skin, gut, and airway in healthy volunteers.

Stage 2 Primary Objective: Determine the combined effects of common vs. pure exposures on the skin, gut, and airway in healthy volunteers.

Endpoints:

Stage 1 Primary Endpoints:

1. Cohort 1 (skin): The primary endpoint for the skin substudy is the skin impedance change response from the common environment (as a log geometric mean ratio [GMR]) minus the mean skin impedance change response from the pure environment (as a log GMR). For each crossover intervention period (common or pure), we measure the GMR as the ratio of the geometric mean (GM) of the average skin impedance measurements at the last day of the inpatient stay over the GM of the average skin impedance measurements at day 0 (baseline).
2. Cohort 2 (GI): The primary endpoint for the GI substudy is analogous to that of the skin substudy, except replacing skin impedance with the Shannon-Weaver diversity index (a measure of metabolic diversity) measured on the gut microbiome.
3. Cohort 3 (airway): The primary endpoint for the airway substudy is the airway maximum change response from the common environment (as the log of the GM of the maximum of the daily change response) minus the airway maximum change response from the pure environment. For each crossover intervention period (common or pure), we measure each individual s daily change response as airway resistance (R5) measured at each day of the inpatient stay over the R5 at day 0 (baseline).

Stage 1 Secondary Endpoints will compare common vs pure crossover period responses as follows:

1. Cohort 1 (skin):

   * Proportion of participants that experience a 30% reduction in skin impedance from admission to any time point during inpatient stay.
   * Change in metabolic functional analysis and/or specific taxa of skin microbiome from admission to last day of the inpatient stay.
   * Change in skin metabolomics by tape strip analysis during study exposure.
2. Cohort 2 (GI):

   * Change in metabolic functional analysis and/or specific taxa of gut microbiome.
   * Change in diversity index, metabolic functional analysis, and/or specific taxa of oral microbiome.
3. Cohort 3 (airway):

   - Increase in R5 from admission to last day of inpatient stay by impulse oscillometry (IOS).
4. All 3 Cohorts:

   * Change in serum and/or intradermal fluid inflammatory markers during study exposure.
   * Change in serum lipopolysaccharides (LPS) and bacterial translocation markers (a marker of GI barrier integrity) during study exposure.
   * Change in quality of life from baseline during exposures to contactants.
   * Change in sense of smell during study exposure.

Stage 2 Endpoint: Based on isolated exposures from single organ systems and randomization design in Stage 1, repeat primary and secondary endpoint responses of Stage 1.

ELIGIBILITY:
* INCLUSION CRITERIA:

To participate in this study, an individual must meet all of the following criteria:

1. Ability to provide informed consent.
2. Age 18-80 years.
3. Agreement to adhere to lifestyle considerations.
4. Ability to exclusively adhere to UPD and MPD during inpatient stay.
5. Ability to speak English.
6. Willing to allow storage of samples and data for future research.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Diagnosis of atopic (physician-diagnosed asthma, AD, food allergy, chronic hives), autoimmune, metabolic, or chronic infectious or inflammatory diseases.
2. Positive Phadiatop test.
3. Current or history of neoplastic disease within 5 years.
4. Use of medication(s) that may affect skin, GI, and/or airway symptoms and may have an effect on skin microbiome, GI microbiome (topical or oral antibiotic use may require 3-6 month delay in enrollment for gut microbiome repopulation, see #8), and/or serum cytokines (other than oral birth control, which is not exclusionary and is allowed during participation provided there is consistence use for 3-6 months prior to enrollment).
5. Current receipt of chemotherapy.
6. HIV, hepatitis B, or hepatitis C infection.
7. Receipt of any vaccine within 1 month prior to enrollment.
8. Receipt of oral antibiotics within 3-6 months prior to enrollment.
9. Use of topical, oral, or parental corticosteroids within 1 month prior to enrollment.
10. Participation in another treatment or intervention study within 3 months prior to enrollment.
11. Currently pregnant or lactating.
12. Currently smoking or vaping.
13. Any other condition or intercurrent illness deemed by the investigators to be of potential risk to the participant or validity of study results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2030-12-30 (Estimated); Study Completion 2031-01-30 (Estimated)

PRIMARY OUTCOMES:
Cohort 1 (skin): The primary endpoint for the skin substudy is the skin impedance change response from the common environment. | Baseline and completion of inpatient stay
  Cohort 1: Determine the effects of common vs. pure exposures on the skin in healthy volunteers.
Cohort 2 (GI): The primary endpoint for the GI substudy is analogous to that of the skin substudy, except replacing skin impedance with the Shannon-Weaver diversity index measured on the gut microbiome that measures metabolic diversity. | Baseline and completion of inpatient stay
  Cohort 2: Determine the effects of common vs. pure exposures on GI tract in healthy volunteers.
Cohort 2 (Airway): The primary endpoint for the airway substudy is the airway maximum change response from the common environment minus the airway maximum change response from the pure environment. | Baseline and completion of inpatient stay
  Cohort 3: Determine the effects of common vs. pure exposures on airway in healthy volunteers
Based on combined exposures from all 3 organ systems and randomization design, repeat primary and secondary endpoint responses of Stage 1. | Baseline and completion of inpatient stay
  Stage 2 Primary Objective: Determine the combined effects of skin, GI, and airway exposures of the respective organ systems in healthy volunteers.

SECONDARY OUTCOMES:
Change metabolic functional analysis, and/or specific taxa of skin microbiome. | Baseline and completion of inpatient stay.
  Compare common vs. pure crossover period responses.
Change in skin metabolomics by tape strip analysis during study exposure. | Baseline and completion of inpatient stay.
  Compare common vs. pure crossover period responses.
Change in metabolic functional analysis, and/or specific taxa of gut microbiome. | Baseline and completion of inpatient stay.
  Compare common vs. pure crossover period responses.
Change in diversity index, metabolic functional analysis, and/or specific taxa of oral microbiome. Perform pair-wise and p-crest analysis. | Baseline and completion of inpatient stay.
  Compare common vs. pure crossover period responses.
Increase in airway resistance (using R5 or R5-R20) from admission to last day (or the maximum of the daily measurements) of inpatient stay by impulse oscillometry (IOS). | Baseline and completion of inpatient stay.
  Compare common vs. pure crossover period responses.
Change in FEV1, FVC using spirometry. | Baseline and last day of inpatient stay.
  Compare common vs. pure crossover period responses.
Change in serum and/or intradermal fluid inflammatory markers. | Baseline and last day of inpatient stay.
  Compare common vs. pure crossover period responses.
Change in serum lipopolysaccharides (LPS) and bacterial translocation markers (a marker of GI barrier integrity). | Baseline and last day of inpatient stay.
  Compare common vs. pure crossover period responses.
Change in quality of life from baseline during exposures to contactants. | Baseline and last day of inpatient stay.
  Compare common vs. pure crossover period responses.

CONTACTS AND LOCATIONS:
Overall Officials: Hirsh D Komarow, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Rinaldi AO, Korsfeldt A, Ward S, Burla D, Dreher A, Gautschi M, Stolpe B, Tan G, Bersuch E, Melin D, Askary Lord N, Grant S, Svedenhag P, Tsekova K, Schmid-Grendelmeier P, Mohrenschlager M, Renner ED, Akdis CA. Electrical impedance spectroscopy for the characterization of skin barrier in atopic dermatitis. Allergy. 2021 Oct;76(10):3066-3079. doi: 10.1111/all.14842. Epub 2021 May 15. PMID 33830511
- [Background] Zeldin J, Chaudhary PP, Spathies J, Yadav M, D'Souza BN, Alishahedani ME, Gough P, Matriz J, Ghio AJ, Li Y, Sun AA, Eichenfield LF, Simpson EL, Myles IA. Exposure to isocyanates predicts atopic dermatitis prevalence and disrupts therapeutic pathways in commensal bacteria. Sci Adv. 2023 Jan 6;9(1):eade8898. doi: 10.1126/sciadv.ade8898. Epub 2023 Jan 6. PMID 36608129
- [Background] Pat Y, Yazici D, D'Avino P, Li M, Ardicli S, Ardicli O, Mitamura Y, Akdis M, Dhir R, Nadeau K, Agache I, Ogulur I, Akdis CA. Recent advances in the epithelial barrier theory. Int Immunol. 2024 Apr 3;36(5):211-222. doi: 10.1093/intimm/dxae002. PMID 38227765
- [Background] Yazici D, Ogulur I, Pat Y, Babayev H, Barletta E, Ardicli S, Bel Imam M, Huang M, Koch J, Li M, Maurer D, Radzikowska U, Satitsuksanoa P, Schneider SR, Sun N, Traidl S, Wallimann A, Wawrocki S, Zhakparov D, Fehr D, Ziadlou R, Mitamura Y, Bruggen MC, van de Veen W, Sokolowska M, Baerenfaller K, Nadeau K, Akdis M, Akdis CA. The epithelial barrier: The gateway to allergic, autoimmune, and metabolic diseases and chronic neuropsychiatric conditions. Semin Immunol. 2023 Nov;70:101846. doi: 10.1016/j.smim.2023.101846. Epub 2023 Oct 4. PMID 37801907
- [Background] Akdis CA. Does the epithelial barrier hypothesis explain the increase in allergy, autoimmunity and other chronic conditions? Nat Rev Immunol. 2021 Nov;21(11):739-751. doi: 10.1038/s41577-021-00538-7. Epub 2021 Apr 12. PMID 33846604
- [Background] Ogulur I, Pat Y, Aydin T, Yazici D, Ruckert B, Peng Y, Kim J, Radzikowska U, Westermann P, Sokolowska M, Dhir R, Akdis M, Nadeau K, Akdis CA. Gut epithelial barrier damage caused by dishwasher detergents and rinse aids. J Allergy Clin Immunol. 2023 Feb;151(2):469-484. doi: 10.1016/j.jaci.2022.10.020. Epub 2022 Dec 1. PMID 36464527
- [Background] Sasaki M, Sundberg M, Frei R, Ferstl R, Heye KN, Willems EP, Akdis CA, Lauener R; CK-CARE Study Group; Roduit C. Electrical impedance spectroscopy detects skin barrier dysfunction in childhood atopic dermatitis. Allergy. 2024 Jan;79(1):142-152. doi: 10.1111/all.15895. Epub 2023 Sep 27. PMID 37753955
- [Background] Yadav M, Chaudhary PP, D'Souza BN, Ratley G, Spathies J, Ganesan S, Zeldin J, Myles IA. Diisocyanates influence models of atopic dermatitis through direct activation of TRPA1. PLoS One. 2023 Mar 6;18(3):e0282569. doi: 10.1371/journal.pone.0282569. eCollection 2023. PMID 36877675
- [Background] Whelan K, Bancil AS, Lindsay JO, Chassaing B. Ultra-processed foods and food additives in gut health and disease. Nat Rev Gastroenterol Hepatol. 2024 Jun;21(6):406-427. doi: 10.1038/s41575-024-00893-5. Epub 2024 Feb 22. PMID 38388570
- [Background] Galant SP, Komarow HD, Shin HW, Siddiqui S, Lipworth BJ. The case for impulse oscillometry in the management of asthma in children and adults. Ann Allergy Asthma Immunol. 2017 Jun;118(6):664-671. doi: 10.1016/j.anai.2017.04.009. PMID 28583260
- [Background] Malvehy J, Hauschild A, Curiel-Lewandrowski C, Mohr P, Hofmann-Wellenhof R, Motley R, Berking C, Grossman D, Paoli J, Loquai C, Olah J, Reinhold U, Wenger H, Dirschka T, Davis S, Henderson C, Rabinovitz H, Welzel J, Schadendorf D, Birgersson U. Clinical performance of the Nevisense system in cutaneous melanoma detection: an international, multicentre, prospective and blinded clinical trial on efficacy and safety. Br J Dermatol. 2014 Nov;171(5):1099-107. doi: 10.1111/bjd.13121. Epub 2014 Oct 19. PMID 24841846
- [Background] Redruello-Requejo M, Del Mar Blaya M, Gonzalez-Reguero D, Robas-Mora M, Arranz-Herrero J, Partearroyo T, Varela-Moreiras G, Penalba-Iglesias D, Jimenez-Gomez P, Reche-Sainz P. Cross-Sectional Comparative Analysis of Gut Microbiota in Spanish Adolescents with Mediterranean and Western Diets. Nutrients. 2025 Jan 22;17(3):388. doi: 10.3390/nu17030388. PMID 39940246
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_002257-I.html